CLINICAL TRIAL: NCT01375348
Title: Cognitive Function in Healthy Volunteers Exposed to Acute Pain Before and After Administration of Remifentanil
Brief Title: Relationship Between Cognitive Function and Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Mech-Sense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: Kogprem
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Cognitive Ability, General
Keywords: Cognitive function; Experimental pain
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Remifentanil (Active Comparator): Investigate the effect of remifentanil on cognitive function in healthy volunteers by use of experimental pain models:
  * tonic muscle pain induced by the tourniquet pain model
  * cognitive tests
  * recording of brain activity by use of 64 channel cap
  Interventions: Drug: Ultiva (remifentanil) or placebo
- Placebo infusion (Placebo Comparator): To blind the study and use as comparator in the investigation of the effect of remifentanil on cognitive function in healthy volunteers by use of experimental pain models:
  * tonic muscle induced pain by the tourniquet pain model
  * cognitive tests
  * brain activity by use of a 64 channel cap
  Interventions: Drug: Ultiva (remifentanil) or placebo

INTERVENTIONS:
Drug: Ultiva (remifentanil) or placebo — 0.1microg/kg/min remifentanil administered as infusion Max infusion time is 20min
  Other Names: Ultiva (remifentanil)

SUMMARY:
Patients with chronic pain can experience considerable changes in their cognitive function such as forgetfulness, increased absentmindedness, confusion etc. Opioids (e.g. morphine and morphine-like analgesics) are often used in treatment of acute and chronic pain and can lead to worsening of the cognitive function. The interaction between pain, treatment and cognitive function is very complex and is far from understood.

The hypothesis of the present study is that by use of experimental pain in healthy volunteers it will be possible to elucidate the interaction between pain, treatment and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men aged 18-65 years
* Normal vision and hearing
* No disease associated with cognitive dysfunction

Exclusion Criteria:

* Allergic to remifentanil or patches
* Any use of pain killers or alcohol 48hours before study start
* Current participation in other clinical studies or participation within the last 14days before study start
* Prescribed medication
* Risk of developing
* Previously alcohol- or drug addict
* MMSE score < 26

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 3 experiments each lasting for about 4-6hours - total duration of study is around 8-9month
  Investigate the relationship between cognitive function and pain and treatment with remifentanil

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, Professor, Principal Investigator — Mech-Sense
Locations (1):
- Mech-Sense, Department of Gastroenterology, Aalborg Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Graversen C, Malver LP, Kurita GP, Staahl C, Christrup LL, Sjogren P, Drewes AM. Altered frequency distribution in the electroencephalogram is correlated to the analgesic effect of remifentanil. Basic Clin Pharmacol Toxicol. 2015 May;116(5):414-22. doi: 10.1111/bcpt.12330. Epub 2014 Oct 21. PMID 25250670